CLINICAL TRIAL: NCT06951399
Title: T-Cell Repertoire Sequencing: Assessing Pembrolizumab Efficacy in Advanced Non-Small Lung Cancer
Brief Title: Tracking T-Cell Responses to Evaluate Pembrolizumab Effectiveness in Advanced Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, ARI RAPHAEL, Head of Translational Oncology, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0026-25-RNC_MK3475-F34
Record Dates: First submitted 2025-04-17; First posted 2025-04-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); NSCLC Stage IV Without EGFR/ALK Mutation; NSCLC Adenocarcinoma
Keywords: metastatic NSCLC adenocarcinoma first-line pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab 200 mg combined with pemetrexed and platinum (cisplatin or carboplatin) (Experimental)
  Interventions: Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: Pembrolizumab (KEYTRUDA®) — IV Pembrolizumab 200 mg combined with pemetrexed and platinum (investigator's choice of cisplatin or carboplatin) every 3 weeks

SUMMARY:
This study includes patients with advanced non-small cell lung cancer (NSCLC) - either unresectable stage III or stage IV adenocarcinoma without actionable driver mutations - who are treated with pembrolizumab in combination with platinum-based doublet chemotherapy, irrespective of PD-L1 expression levels.

The primary objective is to assess treatment response through integration of serial T-cell receptor (TCR) repertoire sequencing (Rep-seq), capturing longitudinal changes in T-cell clonality and diversity. These immune dynamics will be correlated with radiographic response assessed by RECIST 1.1, with the aim of improving the accuracy of response classification, including differentiation between progression, pseudo-progression, and hyperprogression.

Additionally, circulating tumor DNA (ctDNA) levels will be measured longitudinally (pre-treatment and during treatment) to evaluate their potential as a complementary biomarker of disease burden and treatment efficacy in the context of chemo-immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of NSCLC adenocarcinoma stage IV or unresectable stage III.
* Have measurable disease based on RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate organ function.

Exclusion Criteria:

* Aberration in one or more of molecular drivers.
* Has received prior systemic anti-cancer therapy prior to allocation.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in T-cell Receptor (TCR) Repertoire Clonality and Diversity Relative to Disease Response Assessed by RECIST v1.1 | From date of randomization until the end of treatment, defined as a maximum of 35 cycles administered every 3 weeks (up to 2 years), or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first
  TCR sequencing will be performed on peripheral blood samples to assess clonality and diversity metrics. Changes in these metrics will be analyzed relative to clinical disease response evaluated according to RECIST version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Raphael, Principal Investigator — Rabin Medical Center
Locations (1):
- Davidoff Comprehensive Cancer Center, Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428